CLINICAL TRIAL: NCT05397171
Title: A Phase I/IIa First-in-human, Open-label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AZD8853 in Participants With Selected Advanced/Metastatic Solid Tumours
Brief Title: A First-in-human Study to Evaluate the Safety and Tolerability of AZD8853 in Participants With Selected Advanced/Metastatic Solid Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated early as per protocol Section 4.4, based on overall risk-benefit profile observed to date. No safety concerns reported. Only Substudy 1 Part A was started; Parts B & C were not started. Entire Master Protocol was terminated.
Sponsor: AstraZeneca (Industry)
Collaborators: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9450C00001; 2021-005438-41 (EudraCT Number)
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Urinary Bladder Neoplasms; Colorectal Cancer; Carcinoma, Non-Small-Cell Lung
Keywords: AZD8853; Monoclonal antibody; First-in-Human; Non-Small Cell Lung Cancer; Colorectal cancer; Bladder cancer; Urinary Bladder Neoplasms; Growth Differentiation Factor-15 (GDF-15); CD8-Positive T-Lymphocytes; Urothelial Carcinoma; CD8; ⁸⁹Zr-Df-IAB22M2C; PET; Imaging; CD8 + T cells; Zirconium-89 crefmirlimab berdoxam
MeSH Terms: conditions — Urinary Bladder Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Substudy 1:
  * Part A: Part A is an AZD8853 monotherapy dose escalation which may enroll up to 45 participants.
  * Part B: Dose escalation will be followed by Part B, where up to 40 participants will be enrolled to doses determined to be safe during Part A. Additionally, a sub-set of participants will also receive an investigational radiopharmaceutical, Zirconium-89 crefmirlimab berdoxam, to evaluate the presence of CD8+ T cells in and around cancerous tumours.
  * Part C: Part C is an efficacy expansion where up to 80 participants may be enrolled based on doses and indications recommended during Part B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Substudy 1 - Parts A, B, and C (Experimental): * Part A: AZD8853 monotherapy dose escalation
  * Part B1 and Part B2: AZD8853 monotherapy safety expansion at dose levels and indications determined to be safe in Part A
  * Part C1 and Part C2: AZD8853 monotherapy safety and preliminary efficacy expansion at dose levels and indications determined to be safe in Parts A and B
  Interventions: Drug: AZD8853
- Substudy 1 - Parts B1 and B2 with CD8+ PET (Experimental): Sub-set of participants from Parts B1 and B2 will also receive investigational CD8+ T cell targeted radioactive tracer, Zirconium-89 crefmirlimab berdoxam with PET scans
  Interventions: Drug: Zirconium-89 crefmirlimab berdoxam

INTERVENTIONS:
Drug: AZD8853 — Monotherapy given until progressive disease or upon meeting other discontinuation criteria.
  Arms: Substudy 1 - Parts A, B, and C
Drug: Zirconium-89 crefmirlimab berdoxam — CD8+ T cell tracer for positron emission tomography (PET) at two time points in addition to monotherapy AZD8853
  Other Names: 89-Zr-Df-IAB22M2C, 89-Zr-Df-crefmirlimab
  Arms: Substudy 1 - Parts B1 and B2 with CD8+ PET

SUMMARY:
A Phase I/IIa First-in-human, Open-label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AZD8853 in Participants with Selected Advanced/Metastatic Solid Tumours.

DETAILED DESCRIPTION:
This study is evaluating the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of AZD8853 in participants with advanced, unresectable or metastatic Non-Small Cell Lung Cancer (NSCLC), Microsatellite Stable Colorectal Cancer (MSS-CRC), Urothelial Carcinoma (UC).

This is a modular study, that includes a master protocol and Substudies.

Substudy 1 will be conducted in 3 parts - Part A: Dose escalation, Part B: Safety expansion and exploratory CD8+ T cell radiopharmaceutical tracer with PET imaging, and Part C: Efficacy expansion.

ELIGIBILITY:
*Key Inclusion Criteria*

All Substudies:

1. At least one measurable target lesions per RECIST 1.1.
2. Eastern Cooperative Group (ECOG) of 0-1.
3. Life expectancy of ≥ 12 weeks
4. Adequate organ and marrow function as defined in the protocol

Substudy 1:

1. Histologically or cytologically confirmed locally advanced, unresectable or metastatic NSCLC, MSS-CRC, or UC.
2. Documented progression from previous therapy
3. NSCLC:

3.a. At least 1 line of systemic therapy in the advanced / metastatic setting 3.b.Must have received anti-PD-1/anti-PD-L1 agent with or without chemotherapy 3.c. Part B and C: Documented no sensitizing EGFR mutations or ALK fusions/rearrangements

4. MSS-CRC: 4.a. At least 2 prior lines of systemic therapy in the advanced / metastatic setting, including specific therapies defined in the protocol

5. UC: 5.a. At least 1 prior line of systemic therapy in the advanced / metastatic setting, including either a platinum-containing regimen and/or an anti-PD-1 or anti-PD-L1 drug 6. Provision of archival tissue or unstained slides 7. Part B: Willing to provide mandatory biposies at screening and on study 8. Part B-CD8+ PET: At least 1 non-liver lesion suitable for PET imaging

*Key Exclusion Criteria*

All Substudies:

1. Unresolved toxicities ≥ Grade 2 per CTCAE 5.0 from prior therapy, with some exceptions defined in the protocol
2. Symptomatic CNS metastases or leptomeningeal disease
3. Active or ongoing infections, or uncontrolled intercurrent illness as defined in the protocol
4. Active or prior documented autoimmune or inflammatory disorder
5. Body weight loss of > 10% within 30 days of screening visit
6. Type 2 diabetes requiring management by metformin, where metformin cannot be switched to another treatment at least 7 days prior to starting study treatment

Substudy 1:

1. Must not have had a toxicity from a checkpoint inhibitor that lead to permanent discontinuation of immunotherapy
2. Participants with brain metastases, unless treated, asymptomatic, stable, and not requiring treatment

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Research Site, Atlanta, Georgia
  - Research Site, St Louis, Missouri
  - Research Site, Providence, Rhode Island
  - Research Site, Seattle, Washington
- Canada (2):
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9450C00001&attachmentIdentifier=2b97e606-bc6c-470b-b83e-35952d5297d4&fileName=CSR_Synopsis_14_Feb_2024_D9450C00001_Final_AZ_Approved_19th_April_Redacted_PDF-A.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9450C00001&attachmentIdentifier=0ed8fab3-96ef-4144-9fa5-72ab5b1b681c&fileName=D9450C00001_Statistical_Analysis_Plan_28_Jun_2023_final_to_sponsor_Redacted_PDF_A.pdf&versionIdentifier=
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9450C00001&attachmentIdentifier=7b99a193-f200-4969-be95-236c01dd03c7&fileName=D9450C00001_Protocol_amendment-substudy_A2_v3.0_11Apr2022_final_approved_to_sponsor_Redacted_PDF_A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 07 Jun 2022 to 06 Jun 2023 at multiple centers in the United States of America and Canada.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
  Due to early termination of the study, only Part A was started, Parts B & C were not started.
Groups:
- AZD8853 300 mg: Participants with advanced/metastatic solid tumors received AZD8853 300 milligrams (mg) every 3 weeks until progressive disease, unacceptable toxicity, or withdrawal of consent.
- AZD8853 1000 mg: Participants with advanced/metastatic solid tumors received AZD8853 1000 mg every 3 weeks until progressive disease, unacceptable toxicity, or withdrawal of consent.
- AZD8853 3000 mg: Participants with advanced/metastatic solid tumors received AZD8853 3000 mg every 3 weeks until progressive disease, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Started | 3 | 6 | 7
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 7
Not completed — Death | 2 | 3 | 3
Not completed — Study Terminated By Sponsor | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received any amount of investigational product (IP).
Groups:
- AZD8853 300 mg: Participants with advanced/metastatic solid tumors received AZD8853 300 mg every 3 weeks until progressive disease, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg | Total
Number analyzed (Participants) | 3 | 6 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (13.2) | 62.8 (4.2) | 65.1 (7.4) | 63.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data are not reported due to concerns with participant's confidentiality. | 2 | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data are not reported due to concerns with participant's confidentiality. | 4 | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 5 | 5 | 13
  Not reported | 0 | 1 | 1 | 2
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: The safety and tolerability of AZD8853 in participants with selected advanced/metastatic solid tumors was assessed.
  As per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, severity scale ranged from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
  This outcome measure was assessed only for substudy 1 Part A.
Time Frame: From Day 1 up to 90 (±7 days) days after the last dose of AZD8853 (1 Year)
Population: Safety set included all participants who received any amount of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Participants
  Any AE | 3 | 4 | 6
  Any AE possibly related to treatment | 1 | 0 | 2
  Any serious adverse event (SAE) | 1 | 3 | 2
  Any SAE possibly related to treatment | 0 | 0 | 0
  Any SAE with outcome death | 0 | 1 | 0
  Any SAE with outcome death and possibly related to treatment | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 0 | 1 | 0
  Any AE leading to discontinuation of IP and possibly related to treatment | 0 | 0 | 0
  Any AE leading to interruption of IP | 0 | 1 | 1
  Any SAE leading to discontinuation of IP | 0 | 1 | 0
  Any SAE leading to discontinuation of IP and possibly related to treatment (IP) | 0 | 0 | 0
  Any AE of greater than or equal to (>=) CTCAE Grade 3 | 1 | 3 | 4
  Any AE of >= CTCAE Grade 3 possibly related to treatment | 0 | 0 | 0
  Any SAE of >= CTCAE Grade 3 | 1 | 3 | 2
  Any SAE of >= CTCAE Grade 3 possibly related to treatment | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLTs (in dose escalation Parts only) of AZD8853 in participants with selected advanced/metastatic solid tumors was assessed. The DLTs are specific adverse events defined as grade 3 (severe), grade 4 (life-threatening), and grade 5 (death) as per NCI-CTCAE version 5.0 non-hematological toxicity or hematological toxicity. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: From Cycle 1 Day 1 to end of Cycle 1 (21 days)
Population: DLT evaluable set included enrolled participants who completed the DLT evaluation period (defined as 21 days after receiving the first infusion of IP) with at least 75% dosing and had completed safety evaluation requirements during the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR). This outcome measure was assessed only for substudy 1 Part A.
Time Frame: First dose until progression of disease (PD) or last evaluable assessment in the absence of progression (1 Year)
Population: Response evaluable set included all dosed participants who had measurable disease at baseline. Here, "number of participants analyzed" specifies all participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Participants | 0 | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR) at 15 Weeks
Description: Disease control was defined as a best overall response (BOR) of confirmed CR or PR or having stable disease (SD) (without subsequent cancer therapy) maintained for greater than or equal to (>=) 14 weeks (study week 15) from first IP. Disease control rate at study week 15 weeks (DCR-15) was defined as the percentage of participants who had disease control at study week 15 weeks. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: 15 weeks
Population: Response evaluable set included all dosed participants who had measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Participants | 1 | 0 | 1

5. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time from the date of first documented response (which was subsequently confirmed) until the date of documented progression or death in the absence of disease progression. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: First documented response until date of first documented disease progression or study end (1 Year)
Population: Response evaluable set included all dosed participants who had measurable disease at baseline. Only participants in the response evaluable set who had a response were planned to include. However, data was not evaluated for this outcome measure as there were no objective responses available for any participant at any dose level.
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS was defined as the time from the start of study intervention until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from study intervention or received another anti-cancer therapy prior to progression.
  This outcome measure was assessed only for substudy 1 Part A.
Time Frame: First dose until documented disease progression or study end (1 Year)
Population: Safety set included all participants who received any amount of IP.
Measure: Median (Full Range); unit: Months
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Months | 1.31 [1.18 to 3.38] | 1.23 [1.15 to 3.15] | 1.25 [0.95 to 3.29]

7. Secondary Outcome: Percentage Change From Baseline in Tumor Size
Description: Tumor size was the sum of the longest diameters (or short axis measurements for lymph nodes) of the target lesions (TLs). Percentage change in tumor size was determined for participants with measurable disease at baseline. Baseline for Response evaluation criteria in solid tumors (RECIST) version 1.1 was defined as the last evaluable assessment prior to first IP dose. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: Baseline (pre-treatment) up to Week 6 and Week 15
Population: Response evaluable set included all dosed participants who had measurable disease at baseline. Here, "n" (number analyzed in each raw) signifies the participants with available data that were analyzed for each timepoint for this outcome measure.
Measure: Median (Full Range); unit: Percentage change in tumor size
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 6
Percentage change in tumor size
  Week 6 | 10.1 [-0.9 to 16.7] | 10.9 [-0.9 to 41.4] | 14.9 [1.5 to 37.4]
  Week 15: number analyzed (Participants) | 1 | 1 | 2
  Week 15 | 46.5 [46.5 to 46.5] | 5.7 [5.7 to 5.7] | 70.0 [13.2 to 126.7]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the start of treatment until death due to any cause.
  This outcome measure was assessed only for substudy 1 Part A.
Time Frame: First dose until study end (1 Year)
Population: Safety set included all participants who received any amount of IP.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Months | 4.47 [2.92 to NA] — The median and 90% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable at the time of analysis as there was insufficient number of participants with the event of interest (less than 50% for the median estimate) occurred in the study. | 5.45 [2.30 to NA] — The median and 90% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable at the time of analysis as there was insufficient number of participants with the event of interest (less than 50% for the median estimate) occurred in the study. | NA [0.95 to NA] — The median and 90% CI were calculated with the Kaplan Meier process (a process in medical research to measure the proportion of participants surviving for a certain time after receiving treatment) and were non estimable at the time of analysis as there was insufficient number of participants with the event of interest (less than 50% for the median estimate) occurred in the study.

9. Secondary Outcome: Percentage Change in Circulating Tumor Deoxyribonucleic Acid (ctDNA) Levels From Baseline
Description: Change in ctDNA is defined as the percentage change in ctDNA from baseline to each timepoint for the safety population. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: Baseline (pre-treatment), Day 8 of Cycle 1, Days 1 and 8 of Cycle 2, Day 1 of Cycles 3, 4, 5, 7 (each cycle is equal to 21 days)
Population: Safety set included all participants who received any amount of IP. Here, "number of participants analyzed" specifies all participants who were evaluated for this outcome measure and "n" (number analyzed in each raw) signifies the participants with available data that were analyzed for each timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline in ctDNA
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 6
Percentage change from baseline in ctDNA
  Cycle 1 Day 8 | 74.3700 (103.6200) | 30.2546 (98.8909) | 10.7795 (53.1457)
  Cycle 2 Day 1 | 92.1105 (83.4783) | 32.1430 (48.9060) | 20.7386 (78.4507)
  Cycle 2 Day 8: number analyzed (Participants) | 3 | 6 | 3
  Cycle 2 Day 8 | 101.0003 (63.4941) | 84.2143 (101.8080) | 116.3071 (192.7165)
  Cycle 3 Day 1: number analyzed (Participants) | 3 | 4 | 1
  Cycle 3 Day 1 | 64.9807 (22.7578) | 131.5277 (161.3495) | 26.9231 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point.
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 2 | 1
  Cycle 4 Day 1 | -8.3636 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. | 50.2904 (54.8320) | 21.4744 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point.
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 5 Day 1 | 64 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. | 50.4363 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. |
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 7 Day 1 | 67.8182 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. |  |

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of AZD8853
Description: The pharmacokinetic (PK) (Cmax) of AZD8853 in serum when administered in participants with selected advanced/metastatic solid tumors were assessed. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: 0 hour, 15 minutes, 2 hours, 6 hours, 24 hours, 168 hours and 336 hours post EOI of Cycle 1 (each cycle equals to 21 days)
Population: PK analysis set included all participants who received at least one dose of IP with at least one reportable concentration.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (ug/mL)
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Micrograms per milliliter (ug/mL) | 76.70 (3.439) | 339.5 (96.74) | 1121 (225.9)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Last Quantifiable Concentration (AUClast) of AZD8853
Description: The PK (AUClast) of AZD8853 in serum when administered in participants with selected advanced/metastatic solid tumors were assessed. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter (h*ug/mL)
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
Hours*microgram per milliliter (h*ug/mL) | 10080 (1789) | 49210 (12130) | 161100 (43070)

12. Secondary Outcome: Partial Area Under the Plasma Concentration-time Curve From Time 0 to 504 Hours Post Dose (AUC[0-504 Hours]) of AZD8853
Description: The PK (AUC[t1-t2]) of AZD8853 in serum when administered in participants with selected advanced/metastatic solid tumors were assessed. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
h*ug/mL | 11870 (2385) | 57230 (14760) | 189400 (56040)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUCinf) of AZD8853
Description: The PK (AUCinf) of AZD8853 in serum when administered in participants with selected advanced/metastatic solid tumors were assessed. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 7
h*ug/mL | 14580 (4136) | 67480 (18490) | 223700 (79270)

14. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) of AZD8853
Description: The immunogenicity of AZD8853 in participants with selected advanced/metastatic solid tumors were assessed. This outcome measure was assessed only for substudy 1 Part A.
Time Frame: From Day 1 up to 90 (±7 days) days after the last dose of AZD8853 (1 year)
Population: Immunogenicity analysis set included all participants who received at least one dose of IP who have a non-missing baseline ADA result and at least 1 non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 1 | 1 | 0

15. Secondary Outcome: Percentage Change From Baseline in Circulating Growth Differentiation Factor 15 (GDF15) Serum Levels
Description: The pharmacodynamics (PD) activity of AZD8853 by assessment of candidate biomarkers in participants with selected advanced/metastatic solid tumors were assessed. This outcome measure was assessed only for substudy1 Part A.
  End of infusion= EOI; End of treatment= EOT
Time Frame: 0 hours post EOI of Cycle 1 Day 1, Day 1 (Pre-dose) of Cycles 2 and 3 (each cycle equals to 21 days) and 90-days post EOT of 90 days follow-up
Population: PD analysis set included all participants who received at least one dose of IP with at least one reportable concentration. Here, "number of participants analyzed" specifies all participants who were evaluated for this outcome measure and "n" (number analyzed in each raw) signifies the participants with available data that were analyzed for each timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline in GDF15
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
Number analyzed (Participants) | 3 | 6 | 6
Percentage change from baseline in GDF15
  Cycle 1 Day 1: 0 hours post EOI: number analyzed (Participants) | 3 | 4 | 1
  Cycle 1 Day 1: 0 hours post EOI | -97.7850 (0.1917) | -99.2637 (0.1161) | -99.7472 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point.
  Cycle 2 Day 1 (Pre-dose) | 324.2284 (103.7778) | 411.2175 (345.6173) | 165.9668 (82.9703)
  Cycle 3 Day 1 (Pre-dose): number analyzed (Participants) | 1 | 2 | 3
  Cycle 3 Day 1 (Pre-dose) | 636.8307 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. | 770.4598 (520.3336) | 212.5270 (111.5861)
  90 Days Follow-Up: 90 days post EOT: number analyzed (Participants) | 1 | 1 | 1
  90 Days Follow-Up: 90 days post EOT | 2164.2547 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. | 1311.2845 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point. | 2513.913 (NA) — Here, 'NA' indicates that standard deviation was not calculated due to the presence of only one participant at this specific time point.

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to Day -1) up to 90 (±7 days) days after the last dose of AZD8853 (1 Year).
Description: Safety set included all participants who received any amount of IP.
  All the adverse events from Screening till study termination have been presented here before and after receiving treatment.
Arm/Group | AZD8853 300 mg | AZD8853 1000 mg | AZD8853 3000 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/6 | 3/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/6 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 4/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD8853 300 mg (N=3) | AZD8853 1000 mg (N=6) | AZD8853 3000 mg (N=7)
Syncope (Vascular disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD8853 300 mg (N=3) | AZD8853 1000 mg (N=6) | AZD8853 3000 mg (N=7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3
Hypotension (Vascular disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3
Chills (General disorders) | 1 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 2
Haematoma (Vascular disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early as per protocol Section 4.4, based on overall risk-benefit profile observed to date. No safety concerns reported. Only Sub-study 1 Part A was started; Parts B & C were not started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca. Access to this document must be restricted to relevant parties. This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT05397171/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT05397171/SAP_001.pdf